CLINICAL TRIAL: NCT00226174
Title: A Randomized, Placebo-controlled, Double-blind Clinical Trial of Curcuminoids in Oral Lichen Planus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1113-19156-03
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Oral Lichen Planus
Keywords: Curcuminoids; Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Diarylheptanoids

INTERVENTIONS:
Drug: Curcuminoids

SUMMARY:
The purpose of this study is to determine whether curcuminoids are effective in the treatment of oral lichen planus.

DETAILED DESCRIPTION:
Lichen planus is a chronic mucocutaneous, immunologic disease. It can affect the oral mucosa, causing changes that can range from white lace-like patterns on the mucosa, to red atrophic changes to the presence of ulcerations. Symptoms can range from none to severe soreness that greatly interferes with eating. The etiology of lichen planus is not known, and because the tissue damage is mediated by immune cells, lichen planus is considered to be an autoimmune disease. Currently, the most common treatment for oral lichen planus (OLP) is use of systemic and/or topical steroids. These medications though efficacious have side-effects that limit the effectiveness of these treatments.

Tumeric, which comes from the plant curcuma longa, has been used for centuries in Ayurveda (Indian traditional medicine) for its anti-inflammatory properties. In western scientific studies, including invitro studies, animal studies and human studies, components of tumeric called curcuminoids (which include, curcumin (diferuloyl methane), demethoxycurcumin, and bisdemethoxycurcumin) have been found to have anti-inflammatory properties and to be very safe, with few side-effects even at high doses.

The objective of this study is to determine whether curcuminoids, which are safe, non-toxic compounds, can be used to control the signs and symptoms of OLP, a disease which can have serious morbidity, and for which current treatment has significant side-effects. If found to be efficacious, these tumeric extracts will aid patients with OLP in reducing symptoms and therefore the morbidity associated with OLP.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the UCSF oral medicine clinic with oral lichen planus confirmed by biopsy. Patients with either the atrophic or the erosive form of oral lichen planus were eligible.
* Study subjects had to have a symptom score between 3 to 8 at the time of entry into the study. (Range of scale: zero to ten, with zero being no symptoms and ten being the worst imaginable symptoms.)
* Eligible subjects had to have discontinued systemic and/or topical corticosteroids for at least two weeks before entry into the study.

Exclusion Criteria:

* Pregnancy, lactation or unwillingness to use an effective method of contraception. An attempt was to be made to ascertain the date of the last menstrual period among eligible pre-menopausal women. If pregnancy could not be ruled out, a pregnancy test was to be provided to the women before enrollment into the study.
* Patients younger than 21 years of age.
* Patients who could not return for follow-up visits at one week, 4 weeks and 7 weeks after enrollment.
* Patients with a medical contraindication or refusal to take prednisone and or/fluconazole.
* Patients who had a medical contraindication to discontinuation of systemic corticosteroids (eg. those on long term corticosteroid therapy).
* Patients with a history of gastric / duodenal ulcers or gallstones.
* Patients with a history of liver disease.
* Patients on anticoagulants or antiplatelet medications.
* Patients undergoing orthodontic treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Study Completion 2004-09

PRIMARY OUTCOMES:
Change in symptom scores at 7 weeks

SECONDARY OUTCOMES:
Change in clinical signs at one, four and seven weeks
Change in symptom scores at one and four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nita Chainani-Wu, DMD, MPH, MS, Principal Investigator — Assistant Clinical Professor
Locations (1):
- University of California, San Francisco, California, United States

REFERENCES:
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Derived] Chainani-Wu N, Silverman S Jr, Reingold A, Bostrom A, Lozada-Nur F, Weintraub J. Validation of instruments to measure the symptoms and signs of oral lichen planus. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Jan;105(1):51-8. doi: 10.1016/j.tripleo.2007.06.022. PMID 18155609